CLINICAL TRIAL: NCT00315380
Title: Longitudinal Protocol for Eosinophilic Granulomatosis With Polyangiitis
Brief Title: Longitudinal Study for Eosinophilic Granulomatosis With Polyangiitis
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: GlaxoSmithKline (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Peter Merkel, Professor, University of Pennsylvania
Other Study IDs: VCRC5506
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis; Churg-Strauss Syndrome
Keywords: EGPA; CSS
MeSH Terms: conditions — Churg-Strauss Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum and plasma), urine, and DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eosinophilic granulomatosis with polyangiitis (EGPA) is a rare immune system disorder that causes asthma, an excessive number of eosinophils (a type of white blood cell) in the blood, and the inflammation of blood vessels, or vasculitis. In order to properly treat EGPA, it is critical that the level of disease activity can be determined over the course of the disease. The purpose of this study is to determine new biological markers, or biomarkers, that may be used to assess the severity of this disease in people with EGPA.

DETAILED DESCRIPTION:
EGPA, also known as allergic granulomatosis angiitis, is a systemic vasculitis. EGPA is marked by three distinct symptoms: asthma; eosinophilia, evidenced by an excessive number of eosinophils in the blood and tissues; and vasculitis involving the skin, lungs, nerves, kidneys, and other organs. Nerve involvement may also occur in EGPA, causing pain, tingling, numbness, and muscle wasting in the hands and feet. Because EGPA patients may not show any visible signs of active disease, current methods of monitoring disease progression usually represent a period of extended inflammation and disease activity. Thus, patients may go untreated during a period of undetectable disease when damage might be preventable. This study will use novel scientific methods to identify new biomarkers that can be used to monitor disease activity in EGPA patients. These biomarkers may be used to help direct clinical care for EGPA patients and assist in future drug development.

Study visits will occur every 6 months, or annually. Blood and urine collection will occur at every visit. A physical exam and medical and medication history will at every visit; also, participants will be asked to complete several questionnaires to assess disease activity, health status, and tobacco, alcohol, and drug use.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of eosinophilic granulomatosis with polyangiitis are eligible for the study.

Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

- Inability to give informed consent and to sign the consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with eosinophilic granulomatosis with polyangiitis (Churg-Strauss). Enrollment will be sequential and participants will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2006-04; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Discover biomarkers in EGPA capable of measuring disease activity and response to treatment | Study completion

SECONDARY OUTCOMES:
Measure the predictive value of biomarkers for clinical outcome in EGPA | Study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania
Locations (13):
- United States (8):
  - University of California San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
- medius KLINIK KIRCHHEIM, Kirchheim unter Teck, Germany
- AOU Meyer IRCCS, Florence, Italy
- Imperial College Healthcare NHS Trust/ Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heeringa P, Schreiber A, Falk RJ, Jennette JC. Pathogenesis of pulmonary vasculitis. Semin Respir Crit Care Med. 2004 Oct;25(5):465-74. doi: 10.1055/s-2004-836140. PMID 16088492
- [Background] Radice A, Sinico RA. Antineutrophil cytoplasmic antibodies (ANCA). Autoimmunity. 2005 Feb;38(1):93-103. doi: 10.1080/08916930400022673. PMID 15804710
- [Background] Said G, Lacroix C. Primary and secondary vasculitic neuropathy. J Neurol. 2005 Jun;252(6):633-41. doi: 10.1007/s00415-005-0833-9. Epub 2005 Apr 5. PMID 15806339
- [Derived] Doubelt I, Cuthbertson D, Carette S, Khalidi NA, Koening CL, Langford C, McAlear CA, Moreland LW, Monach P, Seo P, Specks U, Warrington KJ, Merkel PA, Pagnoux C. Vitamin D status in ANCA-associated vasculitis. Rheumatol Adv Pract. 2023 Feb 10;7(1):rkad021. doi: 10.1093/rap/rkad021. eCollection 2023. PMID 36874269
- [Derived] Doubelt I, Springer JM, Kermani TA, Sreih AG, Burroughs C, Cuthbertson D, Carette S, Khalidi NA, Koening CL, Langford C, McAlear CA, Moreland LW, Monach PA, Shaw DG, Seo P, Specks U, Warrington KJ, Young K, Merkel PA, Pagnoux C. Self-Reported Data and Physician-Reported Data in Patients With Eosinophilic Granulomatosis With Polyangiitis: Comparative Analysis. Interact J Med Res. 2022 May 25;11(1):e27273. doi: 10.2196/27273. PMID 35612893
- See also: Vasculitis Clinical Research Consortium — http://rarediseasesnetwork.org/cms/vcrc/
- See also: Rare Diseases Clinical Research Consortium — http://rarediseasesnetwork.org/